CLINICAL TRIAL: NCT01069237
Title: Compliance and Contamination in Soft Contact Lens Wearers
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SMA-09-45
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Contact Lens Wear
Keywords: contact lens wear; multi-purpose solution; corneal staining

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OPTI-FREE Replenish: Multi-Purpose Solution for soft contact lenses
  Interventions: Device: OPTI-FREE RepleniSH
- Clear Care: Lens Care Solution for contact lenses
  Interventions: Device: Clear Care

INTERVENTIONS:
Device: OPTI-FREE RepleniSH — Multi-Purpose Solution for soft contact lenses
  Groups: OPTI-FREE Replenish
Device: Clear Care — Lens Care Solution for contact lenses
  Groups: Clear Care

SUMMARY:
The purpose of this study is to assess the lens and lens case microbial colonization associated with marketed care solutions used by experienced soft lens wearers.

DETAILED DESCRIPTION:
The purpose of this study is to assess the lens and lens case microbial colonization associated marketed care solutions used by experienced soft lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Successful contact lens wear on a daily wear basis
* Normal Eyes

Exclusion Criteria:

* Topical ocular medication use
* No active ocular issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Contact Lens Wearers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Microbial colonization on soft contact lenses and lens cases associated with daily lens wear | 2 weeks

SECONDARY OUTCOMES:
Regimen compliance | Baseline, 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, Study Director — Alcon Research